CLINICAL TRIAL: NCT03007446
Title: The Exploratory Study of Conversion Surgery for Apatinib in Combination With Oxaliplatin/S-1(SOX) for Patients With Unresectable Gastric Cancer
Brief Title: The Study of Conversion Surgery for Apatinib in Combination With SOX for Patients With Unresectable Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Lin Chen, Director of the General Surgery Department, Chinese PLA General Hospital, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-BG301
Record Dates: First submitted 2016-12-28; First posted 2017-01-02 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Gastric Cancer
Keywords: Apatinib; SOX; Conversion Surgery; unresectable gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib; Oxaliplatin; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apatinib plus Oxaliplatin/S-1 (Experimental): 1. Apatinib :
     A starting dose of apatinib was administered 500 mg daily on days 1 through 21 of each 3-week cycle.
  2. Oxaliplatin:130 mg/m2，d1，ivgtt，in a 21 day cycle.
  3. S-1:40mg，bid，d1-14，po，in a 21 day cycle.
  Interventions: Drug: Apatinib; Drug: Oxaliplatin; Drug: S-1

INTERVENTIONS:
Drug: Apatinib — Apatinib :A starting dose of apatinib was administered 500 mg daily
  Other Names: Apatinib mesylate tablets
Drug: Oxaliplatin — Oxaliplatin:130 mg/m2，d1，ivgtt，in a 21 day cycle
Drug: S-1 — S-1:40mg，bid，d1-14，po，in a 21 day cycle.

SUMMARY:
This is a Prospective，Single-center，Single-arm，Open-label exploratory clinical trial evaluating the efficacy and safety of Conversion Surgery for Apatinib plus SOX for patients with unresectable gastric cancer.

DETAILED DESCRIPTION:
Gastric cancer is the second most common cause of cancer-related deaths worldwide, and surgical resection during the early stage has improved treatment outcomes.However, many patients are diagnosed with unresectable advanced or metastatic stage disease losing the radical surgery opportunity. Systemic chemotherapy is the leading treatment that prolongs survival times for such patients.

Approximate 20 patients with unresectable gastric cancer will be enrolled in this study,the investigators will evaluate the efficacy and security of Apatinib + SOX(oxaliplatin+S-1) for unresectable gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proved gastric adenocarcinoma;
2. At least a unresectable factor before operation via CT, MRI, or PET-CT: difficult resection of locally advanced gastric cancer(T4b); hepatic metastasis (H1; at most five lesions, total diameter ≤8 cm); Peritoneal metastasis(CY1, P1) ;
3. Definitely diagnosed as unresectable gastric cancer via exploratory laparoscopy or laparotomy;
4. ECOG performance status 0-2;
5. Age 18-70 years old, Life expectancy estimated than 3 months;
6. For results of blood routine test and biochemical tests:

   1. Hgb ≥ 80g/L,
   2. WBC ≥ 4000/mm3,
   3. ANC ≥ 1.5×109/L,
   4. platelets ≥ 80×109/L
   5. ALT and AST ≤ 2.5 x upper normal limit (UNL), and ≤ 5 x UNL（Hematogenous metastases）,
   6. Serum Total bilirubin ≤ 1.5 X UNL,
   7. Serum Creatine ≤ 1.5 x UNL ；
7. Good cardiac function before the recruitment, no seizure of myocardial infarction in past half years, and controllable hypertension and other coronary heart disease;
8. Not concomitant with other uncontrollable benign disease before the recruitment(e.g. the infection in the kidney, lung and liver);
9. informed consent.

Exclusion Criteria:

1. Subjects with poor-controlled arterial hypertension (systolic blood pressure> 140 mmHg and diastolic blood pressure > 90 mm Hg) despite standard medical management; Coronary heart disease greater than Class I; I-level arrhythmia (including QT interval prolongation, for man ≥ 450 ms, for woman ≥ 470 ms) together with Class I cardiac dysfunction; Patients with positive urinary protein;
2. Factors that could have an effect on oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction);
3. Subjects with high gastrointestinal bleeding risk, including the following conditions: local active ulcer lesions with positive fecal occult blood test (++); history of black stool, or vomiting blood in the past 2 months;
4. Contraindications include allergy to apatinib and/or its accessories, active bleeding, intestinal perforation, intestinal obstruction, within 30 days after surgery, drugs with poor-controlled hypertension, Class Ⅲ-Ⅳ cardiac dysfunction （NYHA standard）, severe hepatic and renal dysfunction（level 4）if apatinib use is considered;
5. Abnormal Coagulation (INR>1.5, APTT>1.5 UNL), with tendency of bleed;
6. Pregnant or lactating women;
7. Any other condition that might place the patient at undue risk or preclude a patient from completing the study;
8. Treatment with prior radiotherapy, chemotherapy, Targeted therapy or immunotherapy;
9. Other conditions regimented at investigators' discretion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
reaction rate | 4 months

SECONDARY OUTCOMES:
Objective Response Rate | an expected average of 6 weeks
Disease-free survival | an expected average of 6 weeks
Progression-Free Survival | an expected average of 6 weeks
Overall Survival | 3 years
adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lin Chen, Principal Investigator — the Chinese PLA General Hospital
Locations (1):
- the chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fuchs CS, Tomasek J, Yong CJ, Dumitru F, Passalacqua R, Goswami C, Safran H, Dos Santos LV, Aprile G, Ferry DR, Melichar B, Tehfe M, Topuzov E, Zalcberg JR, Chau I, Campbell W, Sivanandan C, Pikiel J, Koshiji M, Hsu Y, Liepa AM, Gao L, Schwartz JD, Tabernero J; REGARD Trial Investigators. Ramucirumab monotherapy for previously treated advanced gastric or gastro-oesophageal junction adenocarcinoma (REGARD): an international, randomised, multicentre, placebo-controlled, phase 3 trial. Lancet. 2014 Jan 4;383(9911):31-39. doi: 10.1016/S0140-6736(13)61719-5. Epub 2013 Oct 3. PMID 24094768
- [Background] Fukuchi M, Ishiguro T, Ogata K, Suzuki O, Kumagai Y, Ishibashi K, Ishida H, Kuwano H, Mochiki E. Prognostic Role of Conversion Surgery for Unresectable Gastric Cancer. Ann Surg Oncol. 2015 Oct;22(11):3618-24. doi: 10.1245/s10434-015-4422-6. Epub 2015 Feb 7. PMID 25663597
- [Background] Kanda T, Yajima K, Kosugi S, Ishikawa T, Ajioka Y, Hatakeyama K. Gastrectomy as a secondary surgery for stage IV gastric cancer patients who underwent S-1-based chemotherapy: a multi-institute retrospective study. Gastric Cancer. 2012 Jul;15(3):235-44. doi: 10.1007/s10120-011-0100-y. Epub 2011 Oct 28. PMID 22033890
- [Background] Kitayama J, Ishigami H, Yamaguchi H, Yamashita H, Emoto S, Kaisaki S, Watanabe T. Salvage gastrectomy after intravenous and intraperitoneal paclitaxel (PTX) administration with oral S-1 for peritoneal dissemination of advanced gastric cancer with malignant ascites. Ann Surg Oncol. 2014 Feb;21(2):539-46. doi: 10.1245/s10434-013-3208-y. Epub 2013 Aug 22. PMID 23975319
- [Background] Inoue K, Nakane Y, Kogire M, Fujitani K, Kimura Y, Imamura H, Tamura S, Okano S, Kwon AH, Kurokawa Y, Shimokawa T, Takiuchi H, Tsujinaka T, Furukawa H. Phase II trial of preoperative S-1 plus cisplatin followed by surgery for initially unresectable locally advanced gastric cancer. Eur J Surg Oncol. 2012 Feb;38(2):143-9. doi: 10.1016/j.ejso.2011.11.009. Epub 2011 Dec 9. PMID 22154885
- [Background] Ohtsu A, Shah MA, Van Cutsem E, Rha SY, Sawaki A, Park SR, Lim HY, Yamada Y, Wu J, Langer B, Starnawski M, Kang YK. Bevacizumab in combination with chemotherapy as first-line therapy in advanced gastric cancer: a randomized, double-blind, placebo-controlled phase III study. J Clin Oncol. 2011 Oct 20;29(30):3968-76. doi: 10.1200/JCO.2011.36.2236. Epub 2011 Aug 15. PMID 21844504
- [Background] Li J, Qin S, Xu J, Guo W, Xiong J, Bai Y, Sun G, Yang Y, Wang L, Xu N, Cheng Y, Wang Z, Zheng L, Tao M, Zhu X, Ji D, Liu X, Yu H. Apatinib for chemotherapy-refractory advanced metastatic gastric cancer: results from a randomized, placebo-controlled, parallel-arm, phase II trial. J Clin Oncol. 2013 Sep 10;31(26):3219-25. doi: 10.1200/JCO.2013.48.8585. Epub 2013 Aug 5. PMID 23918952